CLINICAL TRIAL: NCT02564809
Title: The Effect of Fit Brains Training on Cognitive Performance in Older Adults
Brief Title: Cognitive Brain Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H14-02438
Record Dates: First submitted 2015-09-01; First posted 2015-10-01 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fit Brains training (Experimental): Both healthy participants and participants with Mild Cognitive Impairment (MCI) will be performing a cognitive training program (Fit Brains training) 6 hours a week for 8 weeks.
  Interventions: Behavioral: Fit Brains Training
- Exercise + Fit Brains training (Experimental): Both healthy participants and participants with Mild Cognitive Impairment (MCI) will be performing a combination of aerobic exercise and a cognitive training program (Fit Brains training) for 6 hours a week over 8 weeks.
  Interventions: Behavioral: Exercise + Fit Brains Training
- Balanced And Tone (Sham Comparator): Both healthy participants and participants with Mild Cognitive Impairment (MCI) will complete 3 weekly training sessions of 1 hour for 8 weeks.
  Interventions: Behavioral: Balanced And Tone

INTERVENTIONS:
Behavioral: Fit Brains Training — These hourly classes will consist of cognitive brain training (Fit Brains by Rosetta Stone) on a mobile device (tablet/iPad). Fit Brains offers 60+ different training games, each targeting one of five cognitive domains - executive functions, memory, concentration/attention, visual-spatial ability, and processing speed. Each game lasts exactly 60 seconds during which individuals aim to answer as many questions correctly. The difficulty of the game increases after each correct answer. Each game has three level of difficulty: 1) novice; 2) intermediate; and 3) advanced.
  Other Names: FBT
  Arms: Fit Brains training
Behavioral: Exercise + Fit Brains Training — These classes combine aerobic training and cognitive training. The classes will consist of a 15-minute walk prior to cognitive brain training (Fit Brains by Rosetta Stone) on a mobile device (tablet/iPad). Fit Brains offers 60+ different training games, each targeting one of five cognitive domains - executive functions, memory, concentration/attention, visual-spatial ability, and processing speed. Each game lasts exactly 60 seconds during which individual aims to answer as many questions correctly. The difficulty of the game increases after each correct answer. Each game has three level of difficulty: 1) novice; 2) intermediate; and 3) advanced.
  Other Names: Ex-FBT
  Arms: Exercise + Fit Brains training
Behavioral: Balanced And Tone — These classes will consist of hourly sham training class, hourly classes of sham exercise (e.g., balance, stretching, range of motion), and hourly educational classes.
  Other Names: BAT
  Arms: Balanced And Tone

SUMMARY:
The investigators will conduct a 8-week proof-of-concept randomized controlled trial to provide preliminary evidence of efficacy of Fit Brains (Rosetta Stone Canada) training -- a mobile cognitive training program -- on cognitive and brain plasticity in older adults. The investigators will also explore whether Fit Brains training paired with a brief bout of exercise would enhance the potential cognitive benefits of Fit Brains. In addition, the investigators will explore the long-term effects of cognitive training by performing a 1-year follow-up measurement (i.e., 1-year after study completion).

DETAILED DESCRIPTION:
This study will look at the effect of FBT on cognitive function in older adults. Additionally, the investigators aim to explore whether a single bout of aerobic exercise prior to Fit Brains training would magnify the training effect on both cognitive and brain outcomes.

Objectives:

1) To compare the effect of Fit Brains training (FBT) and the effect of a single bout of aerobic exercise prior to FBT (Ex-FBT) with a Balanced And Tone (BAT; control) program on cognitive performance in both older adults; 2) To explore the effect of FBT and Ex-FBT with BAT on brain structure and function i; 3) To explore whether the intervention effects (i.e., FBT and Ex-FBT) are moderated by cognitive status (i.e., MCI or not); 4) To explore whether Ex-FBT has additional benefits compared with FBT; and 5) To explore whether potential benefits are maintained at 1-year follow-up.

Research Method:

The investigators will conduct an 8-week proof-of-concept, assessor single-blinded randomized controlled trial (RCT) with 120 older adults (i.e., 40 in each experimental group). A subset of participants will perform MRI scans at baseline and 8-weeks.

To reduce bias, all assessors will be blinded to group allocation of participants. Participants will be randomly assigned to one of the three groups (i.e., FBT, Ex-FBT, or SCT). Participants in the FBT group will be required to attend 3 formal training sessions per week, for 8 weeks, at the Djavad Mowafaghian Centre for Brain Health or the Centre for Hip Health and Mobility. Each session will be for 60 minutes. Additionally, the participants will be asked to complete 3 additional one-hour training sessions at home per week. Thus, the participants will complete a total of 48 hours of cognitive training over 8 weeks.

Participants who are randomized to Ex-FBT will be required to attend 3 formal training sessions per week, for 8 weeks, at the Djavad Mowafaghian Centre for Brain Health or Centre for Hip Health and Mobility. Each session will be for 1 hour. The participants will start the training with a 15-minute walk outside. The 15-minute walk is followed by a 45-minute FBT session (FBT program). Additionally, participants will be asked to complete 3 additional 1-hour training sessions at home (i.e., 15-minute walk followed by 45-minutes of FBT training). Thus, the participants will complete a total of 48 hours of cognitive + walking training over 8 weeks.

Participants who are randomly assigned to the BAT group will be required to attend 3 formal training sessions per week, for 8 weeks, at both the Djavad Mowafaghian Centre for Brain Health and/or the Centre for Hip Health and Mobility. Specifically, the participants will complete a total of 8 hours of sham cognitive training, 8 hours of sham exercise training (Centre for Hip Health and Mobility) and 8 hours of education over the 8 weeks. Thus, the participants will complete a total of 24 hours of sham training over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged between 65 and 85 years
* completed high school education
* live in their own home
* read, write, and speak English with acceptable visual and auditory acuity
* have preserved general cognitive function as indicated by a Mini-Mental State Examination score
* score > 6/8 on the Lawton and Brody Instrumental Activities of Daily Living Scale
* are not expected to start or are stable on a fixed dose of anti-dementia medications (e.g., donepezil, galantamine, etc.) during the 8-week study period
* are able to walk independently;
* are suitable to engage in 15-minutes of brisk walking based on the Physical Activity Readiness Questionnaire; and
* provide a personally signed and dated informed consent document indicating that the individual has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* diagnosed with dementia of any type
* clinically suspected to have neurodegenerative disease as the cause of MCI that is not AD, vascular dementia (VaD), or both (e.g. multiple sclerosis, Parkinson's disease, Huntington's disease, fronto-temporal dementia, etc.)
* have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility, as determined by his/her family physician
* taking medications that may negatively affect cognitive function, such as anticholinergics, including agents with pronounced anticholinergic properties (e.g., amitriptyline), major tranquilizers (i.e., typical and atypical antipsychotics), and anticonvulsants (e.g., gabapentin, valproic acid, etc.)
* planning to participate, or already enrolled in, a concurrent clinical drug trial

Specific exclusion criteria for the MRI subset:

* Participants do not meet the specific scanning requirements of the UBC MRI Research Centre. Specifically, the investigators will exclude anyone with: pacemaker, brain aneurysm clip, cochlear implant, surgery or tattoos within the past 6 weeks, electrical stimulator for nerves or bones, implanted infusion pump, history of any eye injury involving metal fragments, artificial heart valve, orthopedic hardware, other metallic prostheses, coil, catheter or filter in any blood vessel, ear or eye implant, bullets, or other metallic fragments.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in episodic memory as measured with the Rey Auditory Verbal Learning Test (RAVLT) at 8 weeks and 1-year follow-up | Measured at baseline and at program completion (8 weeks), and 1-year follow-up
  Measured by the Rey Auditory Verbal Learning Test (RAVLT)

SECONDARY OUTCOMES:
Change from baseline in response inhibition as measured with the stroop test at 8 weeks and 1-year follow-up | Measured at baseline and at program completion (8 weeks), and 1-year follow-up
  Measured by Standard Neuropsychological Tests and the NIH Toolbox
Change from baseline in set shifting as measured with the Trailmaking A and B test at 8 weeks and 1-year follow-up | Measured at baseline and at program completion (8 weeks), and 1-year follow-up
  Measured by Standard Neuropsychological Tests and the NIH Toolbox
Change from baseline in working memory as measured with the digits forward and backward test at 8 weeks and 1-year follow-up | Measured at baseline and at program completion (8 weeks), and 1-year follow-up
  Measured by Standard Neuropsychological Tests and the NIH Toolbox
Change from baseline in functional capacity as measured by the 6-Minute Walk Test at 8 weeks and 1-year follow-up | Measured at baseline and at program completion (8 weeks), and 1-year follow-up
  Measured by the 6-Minute Walk Test
Change from baseline in mobility as measured by the Short Physical Performance Battery (SPPB) at 8 weeks | Measured at baseline and at program completion (8 weeks).
  Measured by the Short Physical Performance Battery
Change from baseline in brain structure as measured by structural MRI at 8 weeks | Measured at baseline and at program completion (8 weeks).
  Measured by structural MRI
Change from baseline in brain function as measured by resting state functional MRI at 8 weeks | Measured at baseline and at program completion (8 weeks).
  Measured by resting state functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia; John R Best, PhD, Principal Investigator — University of British Columbia; Lindsay S Nagamatsu, PhD, Principal Investigator — University of Western Ontario, Canada; Lisanne F ten Brinke, MSc, Principal Investigator — University of British Columbia; Conny Lin, MsC, Principal Investigator — Rosetta Stone Canada
Locations (1):
- Djavad Mowafaghian Centre for Brain Health & Centre for Hip Health and Mobility, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ten Brinke LF, Best JR, Crockett RA, Liu-Ambrose T. The effects of an 8-week computerized cognitive training program in older adults: a study protocol for a randomized controlled trial. BMC Geriatr. 2018 Jan 30;18(1):31. doi: 10.1186/s12877-018-0730-6. PMID 29378515